CLINICAL TRIAL: NCT01724307
Title: Stimulation of the Cervical Sympathetic Ganglion for Treatment of Asthma.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Parsons (Other)
Responsible Party: Sponsor-Investigator, Jonathan Parsons, M.D., Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011H0009
Record Dates: First submitted 2012-10-09; First posted 2012-11-09 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asthma positive to Methacholine Challenge Testing (Active Comparator): Asthma diagnosis by positive Methacholine Challenge Testing
  Interventions: Procedure: Neurostimulation of stellate ganglion
- Asthma positive to Eucapnic voluntary hyperventilation testing (Active Comparator): Asthma diagnosis by positive Eucapnic voluntary hyperventilation testing
  Interventions: Procedure: Neurostimulation of stellate ganglion

INTERVENTIONS:
Procedure: Neurostimulation of stellate ganglion — An electrical nuerostimulation of the stellate ganglion up to 60 minutes

SUMMARY:
The purpose of this study is to evaluate if stimulating the nerve involved with airway constriction, while undergoing procedures that are known to cause asthma exacerbations, decreases the level of asthma attack experienced.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disorder of the airways characterized by shortness of breath, wheezing, cough, and fatigue. Some people suffer from sudden worsening of asthma symptoms despite being treated with medications. When people have asthma attacks the muscle tissue in the airway contracts causing the airway to narrow and decreasing the ability for the person to breathe.

Neurological pacemakers are FDA approved devices that stimulate nerves in the body and have been used for the treatment of many disorders such as Parkinson's, epilepsy, chronic pain and urinary incontinence. Recent animal studies have shown that stimulating (activating a nerve) the carotid sheath area (located in the neck) can cause the rapid relaxation of the muscles which contract during an asthma attack. This approach has also been successfully used in patients at an emergency room when they came in with a severe asthma attack.

ELIGIBILITY:
Inclusion Criteria:

1. All patients aged 18-70 years of age suffering from mild-to-moderate asthma who have either:

   1. bronchial hyper-responsiveness to MCT
   2. bronchial hyper-responsiveness to EVH testing
2. All patients with documented evidence of a positive MCT or EVH test within 36 months of Visit 1
3. Are capable of reading and understanding questionnaires and providing written informed consent.
4. Are willing and able to adhere to the study visit schedule and other protocol-specified procedures.

Exclusion Criteria:

1. Non-English speaking.
2. Subjects experiencing an exacerbation of asthma within 6 weeks of Visit 1
3. Subjects with a forced expiratory volume (FEV1) ≤ 60% predicted, on spirometry
4. Subjects and medications:

   1. Subjects allergic to methacholine or any other parasympathomimetic agent
   2. Subjects on investigational drugs or participating in interventional research trial(s), 30 days prior to enrollment or during the duration of the study
   3. Subjects currently on β-adrenergic blockers or, a cholinesterase inhibitor
   4. Prior to the administering of the MCT/ EVH test:

   i) use of a short-acting bronchodilator (within 6hrs.) ii) use of a long-acting bronchodilator (within 36hrs.) iii) use of inhaled corticosteroids/ leukotriene modifiers (within 72hrs.) iv) exercise (within 4hrs.)
5. Subject smoking: in the last 6 months or a smoking history of >10 pack-years
6. Subjects who have experienced a febrile illness within 3 weeks of Visit 1
7. Subjects with a history of active poorly controlled epilepsy, cardiovascular disease (esp. with bradycardia), vagotonia, peptic ulcer disease, thyroid disease, or urinary tract obstruction or other chronic ailments that would interfere with the current study
8. Subjects who are pregnant or refuse medically acceptable contraception during the study period
9. Subjects with a history of >3 stellate ganglion block procedures
10. Subjects who have undergone surgical procedures involving the cervical spine
11. Evidence of coagulopathy with abnormal INR, PT/ PTT and platelet count
12. Subjects allergic to lidocaine (Subject may still participate in the study if they agree to the procedure without using the Lidoderm patch)
13. Subjects participating in another interventional research trial
14. Subjects with a condition or compliance issue, which in the investigator's opinion might interfere with participation in the current study
15. Subjects unable or unwilling to provide a written consent to undergo the required testing/ procedures/ physical exam or answer the questionnaires

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Evaluate if neurostimulation of stellate ganglion modulates airway hyperresponsiveness to bronchoprovocation testing. Comparison of FEV1 drop before and after neurostimulation testing will be primary outcome measure | 60 minutes post treatment
  To determine whether neurostimulation of the stellate ganglion modulates airway hyperresponsiveness to bronchoprovocation testing in asthmatics

SECONDARY OUTCOMES:
Evaluate if neurostimulation of the stellate ganglion modulates airway inflammation | 60 minutes post treatment
  To determine whether neurostimulation of the stellate ganglion modulates airway inflammation as measured by exhaled nitric oxide in asthmatics

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Parsons, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States